CLINICAL TRIAL: NCT05938140
Title: Efficiency and Safety of Paxlovid for the Treatment of COVID-19 Patients With Severe Chronic Kidney Disease
Brief Title: Efficiency and Safety of Paxlovid for COVID-19 Patients With Severe Chronic Kidney Disease
Acronym: ESPTCSCKD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Li Zhang, Professor, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChinaPLAGH-2023ESP-CKD
Record Dates: First submitted 2023-06-24; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: COVID-19; Renal Insufficiency, Chronic
MeSH Terms: conditions — COVID-19; Renal Insufficiency, Chronic | interventions — nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paxlovid group (Other): Patients will take Paxlovid.On the first day, Nematavir tablet 300mg/Ritonavir tablet 100mg orally once, then Nematavir tablet 150mg/ Ritonavir tablet 100mg orally once a day for 4 days. Dialysis patients must took the medication after dialysis.
  Interventions: Drug: Nirmatrelvir/ritonavir

INTERVENTIONS:
Drug: Nirmatrelvir/ritonavir — Paxlovid is an oral drug for the treatment of COVID-19. It is suitable for adults with mild to moderate COVID-19 patients with high risk factors for progression to severe disease.
  Other Names: Paxlovid

SUMMARY:
This is a prospective, single-center, open and self-controlled study.The purpose of this study is to evaluate the efficacy and safety of Paxlovid for the treatment of COVID-19 patients with severe chronic kidney disease.

DETAILED DESCRIPTION:
Patients with chronic kidney disease (CKD) have a significantly increased risk of hospitalization or death due to severe COVID-19. A meta-analysis of 348 studies (382,407 COVID-19 and 1,139,979 patients with chronic kidney disease) showed that the incidence of COVID-19 in patients receiving maintenance dialysis was higher than that in CKD patients who did not need renal replacement therapy. The mortality of CKD patients in COVID-19 is higher than that of CKD patients without COVID-19. Another meta-analysis showed that COVID-19 infection was closely related to the mortality of CKD patients. The mortality rate of CKD patients infected with COVID-19 is 5.81 times higher than that of CKD patients not infected with COVID-19.

The severe/critical high-risk groups defined in the novel coronavirus Infection Diagnosis and Treatment Program formulated by the National Health and Wellness Commission include kidney disease and maintenance dialysis patients. It is clearly stated in the treatment plan that adult patients with mild or moderate severity and high risk factors should be treated with antiviral therapy within 5 days of onset.

Naimatevir tablets/ritonavir tablets (Paxlovid) are commonly used antiviral drugs at present, but it is not recommended for patients with severe renal insufficiency at present, mainly because the data of drug metabolism of Naimatevir/Ritonavir in this population are insufficient. Because the efficacy of Naimatevir/Ritonavir in patients with Covid-19 infection is clear, and the small sample of clinical research data of patients with severe renal insufficiency shows that it has a small safety risk, this study intends to carry out the safety and efficacy study of Naimatevir/Ritonavir in CKD5 patients, and at the same time, carry out the pharmacokinetic study to determine whether Naimatevir/Ritonavir can be used in the treatment of CKD5 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Patients with chronic kidney disease above stage 4 (eGFR <30ml/min/1.73m2)
* with positive DNA test or antigen test for COVID-19
* Agree to participate in the study and sign the informed consent form voluntarily

Exclusion Criteria:

* Allergic to any component of nimatevir/ritonavir tablets.
* Drugs that are being or need to be taken that are prohibited to be combined with nimatevir tablets or ritonavir tablets as specified in the instructions (including, but not limited to: methidine, amiodarone, propafenone, quinidine, simvastatin, voriconazole, fusidic acid, rifabutine, rifampicin, colchicine, clozapine, quinoline) thiopine, cisapride, simvastatin, dixima, surazadine, fluoxam, oral midazolam and triazolam etc.)
* Renal transplantation failure is taking an immune agent that namatavir tablets/ritonavir tablets can not combine.
* Severe liver injury (Child-Pugh C) or acute liver failure.
* Critically ill patients requiring ventilator-assisted respiratory support.
* patients who cannot take the whole tablet.
* HIV infection with a viral load greater than 400 copies/ml.
* Suspected or confirmed active systemic infections, other than coronavirus pneumonia, that may have an impact on the evaluation of the study.
* Uremia-related complications include acute heart failure, respiratory failure, severe chronic kidney disease, and cardiovascular disease.
* Patients who are pregnant or are planning a recent pregnancy.
* The researchers didn't consider the patients to be eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Security indexes | Start medication until 14 days
  Adverse and serious adverse events were recorded

SECONDARY OUTCOMES:
SARS-CoV-2 nucleic acid negative transformation time | Start medication until 14 days
  SARS-CoV-2 nucleic acid first positive to negative time.
The proportion of disease that progresses to severe or critical type | Start medication until 14 days
  Severe type refer to any of the following and cannot be explained by other reasons other than Covid-19 infection:
  1. shortness of breath, RR>30 times/minute:
  2. At rest, when inhaling air, the oxygen saturation is less than 93%;
  3. Partial arterial oxygen pressure (Pa02)/ oxygen concentration (Fi02)<300mmHg.
  4. The clinical symptoms are getting worse, and the lung imaging shows that the lesion has obviously progressed more than 50% within 24 ~48 hours.
  Critical type refer to those who meet one of the following conditions:
  1. Respiratory failure occurs and mechanical ventilation is needed;
  2. Shock:
  3. Other organ failure requires ICU monitoring and treatment.
Overall mortality from SARS-CO-2 infection | Start medication until 14 days
  The rate of patients died of Covid-19 infection.
Plotting the concentration-time curve of Paxlovid and its semi-logarithmic curve | Start medication until 14 days
  The concentration-time data of Paxlovid from D1 to D5 were described in a chart, and the dose-time curve and its semi-logarithmic curve were drawn.
PK/PD scatter plots | Start medication until 14 days
  PK/PD scatter plots were established with Paxlovid's plasma concentration as horizontal coordinate and nucleic acid load as vertical coordinate.

CONTACTS AND LOCATIONS:
Overall Officials: Nan Bai, phD, Study Director — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No